CLINICAL TRIAL: NCT06132074
Title: Evaluation of a School Intervention to Influence Knowledge, Attitudes and Behaviour Regarding Consent and Sexual Violence in Adolescents.
Brief Title: Adolescent Consent & Sexual Violence: A School Intervention Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Uppsala University (Other)
Collaborators: Uppsala Tjej- och Transjour (Unknown)
Responsible Party: Principal Investigator, Anna Sarkadi, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-04343-01
Record Dates: First submitted 2023-11-09; First posted 2023-11-15 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Violence Prevention Intervention Evaluation Among Youth

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-arm (Experimental): Immediate scheduling and participation of Uppsala Tjej- och Transjour's intervention.
  Interventions: Behavioral: School sessions on consent, reciprocity and sexual violence
- Wait-list control-arm (Active Comparator): Wait-listed group, will await intervention for 6-8 months. After follow-up measurements, this group will receive the intervention.
  Interventions: Behavioral: School sessions on consent, reciprocity and sexual violence

INTERVENTIONS:
Behavioral: School sessions on consent, reciprocity and sexual violence — The intervention consists of a 120-minute workshop led by a representative from Uppsala Tjej- och Transjour and aims to reduce the vulnerability and prevalence of sexual harassment, sexual violence and to counteract men's violence against women and violence in close relationships by raising awareness among pupils, school staff and guardians about sexual health among young people. The workshop covers areas of consent, reciprocity and sexual violence. The participants will do several valuation based and discussion based exercises regarding these topics and discuss issues, legality, and norms during the time.

SUMMARY:
Since 2015, Uppsala Tjej- och Transjour has run school sessions for secondary school pupils in Uppsala municipality, from year 9 to year 2. The school session is a 120-minute workshop and focuses on increasing knowledge and changing attitudes about consent, reciprocity and sexual violence. The intervention aims to increase participants' knowledge about consent, reciprocity, sex, sexuality and sexual violence in order to create positive attitudinal changes around gender and sexual violence and influence behaviour. The purpose of the study is to evaluate the effect of Uppsala Tjej- och Transjour's school intervention on young people's knowledge, attitudes and behaviour regarding consent, reciprocity and sexual violence. A cluster randomised controlled trial with 16 clusters (89 participants in each cluster) in each arm, a total of 32 clusters. Schools are randomised after baseline measurement to receive the intervention in autumn 2023 or spring 2024 (waiting list). Data collection is done through a questionnaire at two measurement points. A baseline measurement before the intervention (T1) and measurement two (T2) 6 months later. There are still few violence prevention programmes in Sweden that have been evaluated for effectiveness, and several programmes come from the USA. This study is based on a Swedish material and constitutes an important contribution to the development of more effective methods for violence prevention and increased insights into reciprocity and consent.

DETAILED DESCRIPTION:
Background: Young people and LGBTQ+ people are currently, and have long been, over-represented as victims of sexual offences in Sweden. This is clearly illustrated in both statistics from the Swedish National Council for Crime Prevention and in the scientific literature. In order to counteract and prevent violence among young people and boys' violence against girls, the government has created a specific action programme that particularly emphasises preventive measures with the aim of improving knowledge and developing methods. The action programme emphasises the role of schools in working to implement a culture of consent and enhanced violence prevention.

Since 2015, Uppsala Tjej- och Transjour has run school sessions for secondary school pupils in Uppsala municipality, from year 9 to year 2. The schools themselves order the sessions and allocate time for them. The school session is a 120-minute workshop and focuses on increasing knowledge and changing attitudes about consent, reciprocity and sexual violence. The intervention aims to increase participants' knowledge about consent, reciprocity, sex, sexuality and sexual violence in order to create positive attitudinal changes around gender and sexual violence and influence behaviour. The intervention uses awareness-raising materials as well as exercises and group discussion. Uppsala Tjej- och Transjour has a unique position in society where they work closely with young people and the problems that young people experience in everyday life.

Uppsala Tjej- och Transjour, together with Uppsala University, has received funding from the Swedish Gender Equality Agency for an impact evaluation of the school sessions.

Purpose: The purpose of the study is to evaluate the effect of Uppsala Tjej- och Transjour's school intervention on young people's knowledge, attitudes and behaviour regarding consent, reciprocity and sexual violence.

Method: A cluster randomised controlled trial with 16 clusters (89 participants in each cluster) in each arm, a total of 32 clusters. A cluster can be a whole (smaller) school with three parallel classes or a programme in a secondary school with three parallel classes. The schools register as usual, but are randomised after the baseline measurement to receive the intervention in autumn 2023 or spring 2024 (waiting list). Data collection is done through a questionnaire at two measurement points. A baseline measurement before the intervention (T1) and measurement two (T2) 6 months later.

Significance: Violence prevention has previously mainly focused on victims and perpetrators and excluded men from being active participants in prevention programmes. There are still few violence prevention programmes in Sweden that have been evaluated for effectiveness, and several programmes come from the USA. This study is based on a Swedish material and constitutes an important contribution to the development of more effective methods for violence prevention and increased insights into reciprocity and consent.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 15-18 y/o
* Participant goes to a school that is part of the study

Exclusion Criteria:

* Person is under the age of 15 y/o or over the age of 18 y/o
* Person is not enrolled in one of the schools who are part of the study

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge | Baseline, T2 5-6 months later.
  Intervention aims at increasing knowledge about the topics of sexual violence, consent and reciprocity. Participants have answered a survey containing questions on knowledge on these topics which will be followed up 5 months after the intervention has been received and compared with wait-list control-group.
Attitudes | Baseline, T2 5-6 months later.
  Intervention aims at positively effecting attitudes about the topics of sexual violence, consent and reciprocity. Participants have answered a survey containing questions where participants attitudes are measured on these topics. These types of question ask participants to value scenarios or situations presented for them on the topics of the intervention which will be followed up 5 months after the intervention has been received and compared with wait-list control-group.

SECONDARY OUTCOMES:
Behaviour | Baseline, T2 5-6 months later.
  Intervention aims at reducing self-assessed prevalence of different forms of sexual violence. Questions in the survey taken at baseline and in follow-up measurements asks participants questions on their self-assessed experiences with sexual harassment and sexual violence. This will be compared post-intervention with control-group.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sarkadi, Professor, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No